CLINICAL TRIAL: NCT04864886
Title: Metabolic Profiling of Immune Responses in Immune-Mediated Diseases
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000392; 000392-I
Record Dates: First submitted 2021-04-28; First posted 2021-04-29 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01-14

CONDITIONS: Primary Immunodeficiency; Psoriasis; Atopic Dermatitis; Immune-mediated Diseases
Keywords: Primary Immunodeficiency; Psoriasis; Atopic Dermatitis; pathways; Natural History
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Psoriasis; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy volunteers: Control group
- Patients with atopic dermatitis: Physician-diagnosed atopic dermatitis
- Patients with primary immunodeficiency: Confirmed by genetic diagnosis or suspected by genetic variant of unconfirmed significance and a history consistent with immunodeficiency
- Patients with psoriasis: Physician-diagnosed psoriasis

SUMMARY:
Background:

The immune system is the part of the body that fights infection. Some people have immune deficiencies that cause skin rashes, make them get sick often with infections, or make it difficult for their skin to heal. Researchers want to learn more to better treat conditions that affect immune response.

Objective:

To learn about how the immune system and skin healing are related to each other.

Eligibility:

People ages 18-75 with primary immune deficiency, eczema, or psoriasis. Healthy volunteers are also needed.

Design:

Participants will be screened with a medical and medicine history and a physical exam. They may take a pregnancy test.

Participants will discuss the medicines or supplements they take as well as skin products they use, such as soaps and lotions.

Participants will have up to 4 skin biopsies taken from the forearm. A needle will inject an anesthetic into the skin where the biopsy will be done. A sharp tool that looks like a tiny cookie cutter will be used to remove a round plug of skin a bit smaller than the tip of a pencil.

Participants will give at least 1 blood sample.

Participants may have optional skin swab collection. A cotton swab will be used to swab the skin on the arm.

Participants may have optional skin tape collection. A sticky strip of tape will be placed on the arm and then removed.

Participants may give leftover samples taken as part of their regular medical care.

Participation will last for about 4 days. Participants will have 2 visits that each last about 1 hour. They may be asked to repeat the study in the future.

DETAILED DESCRIPTION:
Study Description:

This is an exploratory sample collection study enrolling adult healthy volunteers and patients with immune-mediated diseases to elucidate the metabolic signatures associated with immune-mediated diseases. We hypothesize that activation of, and responses to, specific immune pathways will require metabolic changes within cells, serum, and skin.

Following screening and baseline procedures, including blood draw, participants who are able to attend onsite visits will undergo skin biopsies. The skin biopsies will involve up to 4 biopsies: 2 initial punch biopsies 2 mm in diameter, optionally followed by 1 or 2 punch biopsies 3 (+/-10) days later using a 3-mm punch to encompass the initial biopsy site(s), capturing the tissue at 3-14 days of healing. There will be an option for blister induction to maximize keratinocyte collection. Blister induction involves creating 8 blisters on the forearm and removing the tops of the blisters for primary cell culture derivation. In addition, skin swabs and tape strips may be collected to assess for microbial or host markers of epithelial repair. Peripheral blood and functional signatures will be collected with the initial and follow-up biopsies to compare metabolic and functional signatures in peripheral blood cells and serum with those in the skin. Urine may be collected in order to detect metabolites that are not as easily detected in the blood. After day 0 (or 3-14, if the participant has that optional visit), participation in the study will be complete. At-home participants who cannot attend onsite visits may enroll for survey

data collection and optional at-home sample collection (with at least one sample type required). Exposome data will be collected to assess how environmental, occupational, and dietary exposures associate with the results.

Samples and data will be stored for future research use.

Objectives:

Primary Objectives:

1. Evaluate metabolic profiles in immune activation associated with known or suspected immune-mediated disorders.
2. Determine whether there are abnormalities in specific tissue repair pathways, such as epithelial to mesenchymal transition (EMT), that are associated with immune-mediated disorders.

Secondary Objectives:

Not applicable.

Exploratory Objective:

Evaluate how metabolic profiles in immune activation vary with differing occupational, environmental, and/or dietary exposures.

Endpoints:

Primary Endpoints:

1. Fold differences in metabolic pathways associated with immune pathways.
2. Fold differences in metabolic pathways related to wound healing.
3. Change in relative abundance of microbial skin taxa and/or skin metabolites associated with wound healing or immune-mediated disorders.

Secondary Endpoints:

Not applicable.

Exploratory Endpoints:

1. Association between fold differences in metabolic pathways associated with immune pathways and environmental, occupational, and/or dietary exposures.
2. Association between fold differences in metabolic pathways related to wound healing and environmental, occupational, and/or dietary exposures.
3. Association between change in relative abundance of microbial skin taxa and/or skin metabolites associated with wound healing or immune-mediated disorders and environmental, occupational, and/or dietary exposures.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Meets one of the following:

   1. Has documentation of PID confirmed by genetic evaluation demonstrating a deleterious variant in the gene (or genes) known to be associated with immune deficiency (confirmed PID); or
   2. Has documented variant of undetermined significance in a gene (or genes) that is predicted to be deleterious in immune function by the investigators OR a clinical history of infections which are more frequent, more chronic, or more severe than normal (suspected PID); or
   3. Has physician-diagnosed psoriasis; or
   4. Has physician-diagnosed AD; or
   5. Does not have clinically apparent evidence of any monogenic or digenic immune defect, AD, or psoriasis (healthy volunteers).
2. Aged 18 to 75 years.
3. Willing to allow storage of blood, biopsy tissue, bacterial and fungal cultures, and any other samples collected for future research.
4. Able to provide informed consent.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Current or prior (within 3 months) anticoagulant or anti-platelet therapy (other than aspirin or non-steroidal anti-inflammatory drugs).
2. Current or prior (within 3 months) use of immunomodulatory drugs (eg, chemotherapy, steroids), except if approved by the principal investigator.
3. History of keloid formation.
4. Pregnancy, lactating, or breastfeeding.
5. Any condition that, in the opinion of the investigator, contraindicates participation in the study.

Co-enrollment guidelines: Participants may be co-enrolled in other studies; however, study staff should be notified of co-enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers will be recruited through the Clinical Research Volunteer Program. We anticipate that most patient participants will be existing CC participants referred from ongoing NIH protocols;they may also be self-referred through their own initiative or referred by outside physicians.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in relative abundance of microbial skin taxa and/or skin metabolites associated with wound healing or immune mediated disorders. | Throughout study
  Determine whether there are abnormalities in specific tissue repair pathways, such as epithelial to mesenchymal transition (EMT) are associated with immune-mediated disorders.
Fold difference in metabolic pathways associated with immune pathways. | Throughout study
  Evaluate metabolic profiles in immune activation associated with known or suspected immune-mediated disorders.
Fold differences in metabolic pathways related to wound healing. | Throughout study
  Determine whether there are abnormalities in specific tissue repair pathways, such as epithelial to mesenchymal transition (EMT) are associated with immune-mediated disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Myles, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] McCann KJ, Yadav M, Alishahedani ME, Freeman AF, Myles IA. Differential responses to folic acid in an established keloid fibroblast cell line are mediated by JAK1/2 and STAT3. PLoS One. 2021 Mar 4;16(3):e0248011. doi: 10.1371/journal.pone.0248011. eCollection 2021. PMID 33662027
- [Background] Dmitrieva NI, Walts AD, Nguyen DP, Grubb A, Zhang X, Wang X, Ping X, Jin H, Yu Z, Yu ZX, Yang D, Schwartzbeck R, Dalgard CL, Kozel BA, Levin MD, Knutsen RH, Liu D, Milner JD, Lopez DB, O'Connell MP, Lee CR, Myles IA, Hsu AP, Freeman AF, Holland SM, Chen G, Boehm M. Impaired angiogenesis and extracellular matrix metabolism in autosomal-dominant hyper-IgE syndrome. J Clin Invest. 2020 Aug 3;130(8):4167-4181. doi: 10.1172/JCI135490. PMID 32369445
- [Background] Myles IA, Castillo CR, Barbian KD, Kanakabandi K, Virtaneva K, Fitzmeyer E, Paneru M, Otaizo-Carrasquero F, Myers TG, Markowitz TE, Moore IN, Liu X, Ferrer M, Sakamachi Y, Garantziotis S, Swamydas M, Lionakis MS, Anderson ED, Earland NJ, Ganesan S, Sun AA, Bergerson JRE, Silverman RA, Petersen M, Martens CA, Datta SK. Therapeutic responses to Roseomonas mucosa in atopic dermatitis may involve lipid-mediated TNF-related epithelial repair. Sci Transl Med. 2020 Sep 9;12(560):eaaz8631. doi: 10.1126/scitranslmed.aaz8631. PMID 32908007
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000392-I.html